CLINICAL TRIAL: NCT07287839
Title: Phase-2 Trial of Parcel-guided rTMS for Major Depressive Disorder
Brief Title: Parcel-guided rTMS for Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: Columbia University Irving Medical Center, New York, NY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTMSP2
Record Dates: First submitted 2025-12-13; First posted 2025-12-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: rTMS; TMS; parcel-guided; beam-F3
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard rTMS (Active Comparator): rTMS using standard targeting (Beam-F3) will be delivered
  Interventions: Device: Accelerated rTMS
- Parcel-guided rTMS (Experimental): rTMS will be delivered using brain-surface parcellation targeting
  Interventions: Device: Parcel-guided Accelerated rTMS

INTERVENTIONS:
Device: Accelerated rTMS — rTMS targeting will be done using the standard Beam-F3 targeting method. Treatment will be delivered in an accelerated schedule with 50 treatment session over 5 days.
  Arms: Standard rTMS
Device: Parcel-guided Accelerated rTMS — rTMS targeting will be done using brain surface parcellation. Treatment will be delivered in an accelerated schedule with 50 treatment sessions over 5 days.
  Arms: Parcel-guided rTMS

SUMMARY:
Study comparing standard repetitive transcranial magnetic stimulation (rTMS) for Depression to a novel targeting approach using brain surface parcellation to locate a specific brain target.

DETAILED DESCRIPTION:
Standard rTMS treatment often uses the "Beam-F3" targeting approach to locate a brain region known as the left dorsolateral prefrontal cortex (lDLPFC). However, Beam-F3 does not take into account interindividual variation in brain anatomy. Researchers as Columbia University have found a more accurate and personalized approach that uses MRI-based brain surface parcellation to locate the specific subregion of the lDLPFC most ideal for rTMS treatment. Our study is comparing standard rTMS (Beam-F3) to parcel-guided rTMS for patients with treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of major depressive disorder confirmed using the Mini International Neuropsychiatric Interview (MINI30) Axis 1 and mood modules
* Treatment-resistant MDD during the current major depressive episode documented in the MGH Antidepressant Treatment History Questionnaire (ATRQ31), which will be defined as being non-responders (less than 50% of symptom improvement) to two or more depression treatment trials of adequate dose and duration as defined by the MGH ATRQ.
* At least moderate depression severity, operationalized as Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 20

Exclusion Criteria:

* Ever met criteria for a psychotic disorder (Sz, SzAff, Bipolar disorder)
* Anorexia nervosa or bulimia nervosa within the last year
* Unstable medical condition by history, physical exam or laboratory results
* Currently pregnant or breastfeeding women; fecund women not using adequate contraceptive methods or with plan to become pregnant
* Contraindications to MRI (based on metal screening form)
* Meets criteria for claustrophobia
* Recent drug or alcohol use disorder with DSM-5 specifier of moderate or severe within 6 months, or mild within 2 months; or lifetime history of IV drug use A- ctively suicidal, as defined by expressive ideation with a plan or with suicidal ideation that requires immediate medical or treatment intervention.
* Neurological or neuromuscular disorder
* Requires medications for a general medical condition that contraindicate the TMS treatment
* Prior non-response to ECT, vagal nerve stimulation (VNS) or deep brain stimulation (DBS)
* History of ketamine treatment within 6 months
* History of monoamine oxidase inhibitor (MAOI) within the past month
* Lacks capacity to consent
* Taking medications that increase the risk of seizures.
* For patients on permitted concomitant psychotropic agents (antidepressants, anticonvulsants, benzodiazepines, hypnotics, opiates, triiodothyronine (T3), modafinil, psychostimulants, buspirone, melatonin, omega-3 fatty acids, folate, l-methylfolate, s-adenosyl methionine, lithium) dosing must be stable for at least four weeks prior to study entry and patients must agree to continue at the same dose during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline and at end of Week 1
  Depression severity scale with a score ranging from 0 to 60 where a higher score indicates greater severity of symptoms.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale Anxiety Somatization Subscale (HAMD-AS) | Baseline and at Week 1
  six-item subscale of psychiatric disorder severity where a score is given between 0 and 18 and a higher score indicates greater severity of symptoms
Side-effect form (SEF) | Daily from Baseline until Week 1
  Clinician-rated simple form to document the onset, course, severity, and causality of adverse events
Columbia suicide severity rating scale (C-SSRS) | Baseline and Week 1
  Rating scale for suicidal ideation with scores ranging from 0 to 5 where a higher score indicates greater severity of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Datta, PhD, Principal Investigator — Soterix Medical, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno-Ortega M, Kangarlu A, Lee S, Perera T, Kangarlu J, Palomo T, Glasser MF, Javitt DC. Parcel-guided rTMS for depression. Transl Psychiatry. 2020 Aug 12;10(1):283. doi: 10.1038/s41398-020-00970-8. PMID 32788580